CLINICAL TRIAL: NCT06163404
Title: A Prospective, Multi-Center, Open-Label Study to Evaluate the Safety and Effectiveness of the Spirair Implant for Correction of Cartilaginous Nasal Septal Deviation
Brief Title: Open-Label Study to Evaluate the Safety and Effectiveness of the Spirair Implant
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spirair, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-002
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Nasal Septal Deviation; Nasal Airway Obstruction
Keywords: NAO; Septal Deviation; Mobile Cartilaginous Nasal Septal Deviation
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Intervention Model Description: Device: Spirair NSD system for minimally invasive correction of nasal septal deviation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Investigational Device (Experimental): Treatment with the Spirair Septal correction device and delivery system for correction of cartilaginous nasal septal deviation.
  Interventions: Device: Implantation of Spirair Nasal Device using the Spirair delivery system.

INTERVENTIONS:
Device: Implantation of Spirair Nasal Device using the Spirair delivery system. — The Spirair implant is designed to acutely correct cartilaginous septal deviation and maintain the cartilage in a corrected position for a duration sufficient to allow for cartilaginous remodeling.
  Other Names: SeptAlign

SUMMARY:
Pilot study of bioabsorbable implant and delivery device for correction of septal deviation.

DETAILED DESCRIPTION:
To evaluate the safety and effectiveness of the Spirair Implant as a primary treatment for correction of cartilaginous nasal septal deviation.

ELIGIBILITY:
Inclusion Criteria:

* ≥21 to ≤ 70 years of age at time of consent
* Seeking treatment for nasal airway obstruction (NAO) symptoms due primarily to cartilaginous nasal septal deviation
* Willing to undergo a nasal implant procedure
* NOSE score ≥30 at Baseline Visit
* Non-calcified, mobile cartilaginous nasal septal deviation

Exclusion Criteria:

* Target nasal septal deviation that is calcified or non-mobile
* Previous septoplasty or rhinoplasty
* Having a concurrent ENT procedure, other than turbinate reduction
* Saddle nose deformity
* Congenital nasal defect
* Documented evidence that middle meatus is not visualized on endoscopic exam due to severe septal deviation
* Turbinate reduction within the past six (6) months
* Permanent implant or dilator in the nose
* History of nasal vasculitis, unhealed wounds, cartilaginous nasal septal perforation or mucosal irregularities
* Active infection at the impllantation site e.g., folliculitis
* Current or chronic systemic steroid and/or has had radiation exposure or active chemotherapy in the treatment area
* Polyps or pathology, other than turbinate hypertrophy, that may be primary contributor to airway obstruction, in the opinion of the Investigator
* History of a significant bleeding disorder(s) and or taking current prescription blood thinner medication
* Hypersensitivity to any investigational device materials inclusing known or suspected allergy to poly(dioxanone) (PDO) or other bioabsorbable materials
* Major medical condition that could affect quality of life or wound healing and influence the results of the study (e.g., poorly controlled diabetes, HIV or other immunosuppressive conditions, active malignancy in the past 5 years, acute MI, CVA, etc.)
* Active smoker or history of tobacco or tobacco-related product use within the past 1 year
* Documented evidence of a history (e.g., liver testing) of drug/alcohol abuse within 12 months of enrollment
* Females of child-bearing potential who are either pregnant or breastfeeding or plan to become pregnant during the course of the study
* Currently participating, or plans to enroll in another clinical trial during this study or undergo another nasal septal treatment during study participation
* History of non-compliance with medical treatment or clinical trial participation
* Subject is physically or mentally compromised (e.g., currently being treated for a psychiatric disorder, senile dementia, Alzheimer's disease, etc.), to the extent that the Investigator determines the subject to be unable or unlikely to comply with protocol required follow-up
* Any comorbidity or condition that renders the patient a poor surgical candidate as determined by the Investigator
* The subject is receiving prescription narcotic pain medication
* The subject's condition represents a worker's compensation case
* Symptoms of an upper respiratory infection e.g., runny nose, sneezing
* History of untreated or inadequately controlled rhinitis (allergic and/or nonallergic)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 3 Months
  Percent change in Nasal Obstruction Septoplasty Effectiveness scale (NOSE) improvement at Month 3 compared to baseline.
Primary Safety Endpoint | 3 Months
  Incidence of Serious Adverse Device Effects (SADEs), through Month 3.

SECONDARY OUTCOMES:
Secondary Endpoint - 1 | 12 Months
  Mean change in Nasal Obstruction Septoplasty Effectiveness Scale (NOSE) from baseline.
Secondary Endpoint - 2 | 12 Months
  Change in Sino-Nasal Outcomes Test (SNOT-22) from baseline.
Secondary Endpoint - 3 | 12 Months
  Change in Euro QOL Five Dimensions Questionnaire (EQ-5D-5L) from baseline.
Secondary Endpoint - 4 | 12 Months
  Change in Nasal Airway Obstruction (NAO) Visual Analog Scale (VAS) from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon McCutcheon, MD, Study Director — Spirair, CMO
Locations (8):
- United States (8):
  - Alabama Nasal and Sinus Center, Birmingham, Alabama
  - Breathe Clear Institute, Torrance, California
  - Kentuckiana Ear, Nose & Throat, Louisville, Kentucky
  - Sinus and Nasal Specialists of LA, Baton Rouge, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Albany ENT & Allergy Services, PC, Albany, New York
  - Specialty Physicians, Bethlehem, Pennsylvania
  - Ear Nose Throat & Allergy Associates, Puyallup, Washington

IPD SHARING:
Plan to Share IPD: No